CLINICAL TRIAL: NCT05853731
Title: The Feasibility of Using Green Light Phototherapy for the Management of Acute Postoperative Pain
Brief Title: The Effect of Light Therapy on Post-Surgical Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to lack of resources
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sean P. Kiley, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-011669
Record Dates: First submitted 2023-04-29; First posted 2023-05-11 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Intensive Care Unit; Cardiac Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Green light therapy group (Experimental): Subjects in the intensive care unit (ICU) setting after cardiac surgery will have green light therapy via green light emitting diode (GLED) for the duration of the ICU stay or up to 1 week.
  Interventions: Device: Green light emitting diode
- Placebo Group (Placebo Comparator): Subjects in the intensive care unit (ICU) setting after cardiac surgery will have filtered white light emitting diodes (WLED) as a placebo for the duration of the ICU stay or up to 1 week.
  Interventions: Device: White light emitting diode

INTERVENTIONS:
Device: Green light emitting diode — Green light therapy via light emitting diode (LED) in the 520 nanometers (nm) range at 4 lux intensity for up to 5 hours per day, as tolerated.
  Other Names: GLED
  Arms: Green light therapy group
Device: White light emitting diode — Filtered white light via light emitting diode (LED) displayed for up to 5 hours per day, as tolerated
  Other Names: WLED
  Arms: Placebo Group

SUMMARY:
Researchers aim to demonstrate that the use of phototherapy is feasible and may reduce acute postoperative pain based on recent literature. The primary objective is to demonstrate that displaying light-emitting diodes [LED] can be achieved in the ICU setting in after cardiac surgery.

DETAILED DESCRIPTION:
The primary aim of this study to determine whether or not green light phototherapy is feasible after cardiac surgery.

Patients that will be undergoing heart surgery will be recruited to the study. After surgery they will be exposed to either green or white LEDs for up to 5 hours per day and up to one week after surgery.

After their exposure to light therapy, a survey will be given to the patient which will ask questions regarding tolerance of the therapy. A survey will also be given to the staff which will query whether or not the therapy was an impediment to workflow. In addition, the medical record will be reviewed to assess opiate usage in each group as an exploratory aim which may suggest differences in pain experiences.

ELIGIBILITY:
Inclusion Criteria:

- Status post heart surgery and are admitted in the ICU at Mayo Clinic, Florida.

Exclusion Criteria:

* Patient with color blindness and/or untreated cataracts.
* Patients who are hemodynamically unstable.
* Patients with dementia/delirium.
* Pregnancy.
* Patient is unwilling to participate or provide informed consent.
* High baseline narcotic baseline requirements that would skew the baseline impact on post-op opiate pain requirements.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in postoperative pain | Baseline, 1 week
  Measured pain numeric rating scale from 0-10, where 0 was no pain and 10 was the worst pain imaginable. In this scale, a higher number indicates worse outcome and lower number indicates better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Kiley, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials